CLINICAL TRIAL: NCT03850444
Title: A Randomized, Open Label, Phase III Study of Overall Survival Comparing Pembrolizumab (MK-3475) Versus Platinum Based Chemotherapy in Treatment Naïve Subjects With PD-L1 Positive Advanced or Metastatic Non-Small Cell Lung Cancer (Keynote 042)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Platinum-Based Chemotherapy for Participants With Programmed Cell Death-Ligand 1 (PD-L1)-Positive Advanced or Metastatic Non-Small Cell Lung Cancer (MK-3475-042/KEYNOTE-042)-China Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-042 China Extension; 152877 (Other: JAPIC-CTI); MK-3475-042 (Other: Merck); KEYNOTE-042 (Other: Merck)
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Results first posted 2019-08-26 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Programmed Cell Death 1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL 1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL 2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg by IV infusion on Day 1 every 3 weeks (Q3W) for a maximum of 35 cycles (21-day cycles). Participants who stop the initial course of pembrolizumab due to complete response or complete the initial course of pembrolizumab and have stable disease, but progress after discontinuation, are eligible for a second course of pembrolizumab for up to an additional 1 year (17 additional 21-day cycles).
  Interventions: Biological: pembrolizumab
- SOC Treatment (Active Comparator): Participants receive carboplatin at target dose Area Under the Curve (AUC 5) (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + paclitaxel 200 mg/m^2 by IV infusion on Day 1 Q3W for a maximum of 6 cycles (21-day cycles) OR carboplatin target dose AUC 5 (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + pemetrexed 500 mg/m^2 by IV infusion on Day 1 Q3W for a maximum of 6 cycles (21-day cycles). Participants with non-squamous histologies receive optional additional maintenance treatment with pemetrexed 500 mg/m^2 by IV infusion on Day 1 Q3W.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: pemetrexed

INTERVENTIONS:
Biological: pembrolizumab
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab
Drug: carboplatin
  Other Names: PARAPLATIN®
  Arms: SOC Treatment
Drug: paclitaxel
  Other Names: TAXOL®
  Arms: SOC Treatment
Drug: pemetrexed
  Other Names: ALIMTA®
  Arms: SOC Treatment

SUMMARY:
In the China extension study, Chinese participants with programmed cell death ligand 1 (PD-L1)-positive non-small cell lung cancer (NSCLC) will be randomized to receive single agent pembrolizumab for up to 35 treatments or standard of care (SOC) platinum-based chemotherapy (carboplatin + paclitaxel or carboplatin + pemetrexed for 4 to 6 21-day cycles). Chinese participants in the platinum-based chemotherapy arms with non-squamous tumor histologies may receive pemetrexed maintenance therapy after the 4 to 6 cycles of chemotherapy. The primary extension study hypothesis is that pembrolizumab prolongs overall survival (OS) compared to SOC chemotherapy in Chinese participants.

DETAILED DESCRIPTION:
The China extension study enrolled 262 participants. Of the 262 total participants enrolled, 92 were also previously enrolled in the global study for MK-3475-042 (NCT02220894).

ELIGIBILITY:
Inclusion criteria:

* Histologically- or cytologically-confirmed diagnosis of advanced or metastatic NSCLC
* PD-L1 positive tumor
* Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Life expectancy of at least 3 months
* No prior systemic chemotherapy for the treatment of the participant's advanced or metastatic disease (treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as completed at least 6 months prior to diagnosis of advanced or metastatic disease)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ function
* No prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or in situ cancer, or has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy
* Submission of formalin-fixed diagnostic tumor tissue (in the case of participants having received adjuvant systemic therapy, the tissue should be taken after completion of this therapy)
* Female participants of childbearing potential must have a negative urine or serum pregnancy test and must be willing to use two adequate barrier methods of contraception or a barrier method plus a hormonal method starting with the screening visit through 120 days after the last dose of pembrolizumab or 180 days after the last dose of chemotherapeutic agents used in the study
* Male participants with a female partner(s) of childbearing potential must be willing to use two adequate barrier methods of contraception from screening through 120 days after the last dose of pembrolizumab or 180 days after the last dose of chemotherapeutic agents used in the study

Exclusion criteria:

* Epidermal growth factor receptor (EGFR)-sensitizing mutation and/or is echinoderm microtubule-associated protein-like 4 (EML4) gene/anaplastic lymphoma kinase (ALK) gene fusion positive
* Currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study therapy
* No tumor specimen evaluable for PD-L1 expression by the central study laboratory
* Squamous histology and received carboplatin in combination with paclitaxel in the adjuvant setting
* Is receiving systemic steroid therapy ≤3 days prior to the first dose of study therapy or receiving any other form of immunosuppressive medication with the exception of daily steroid replacement therapy
* The NSCLC can be treated with curative intent with either surgical resection and/or chemoradiation
* Expected to require any other form of systemic or localized antineoplastic therapy while on study
* Any prior systemic cytotoxic chemotherapy, biological therapy or major surgery within 3 weeks of the first dose of study therapy; received lung radiation therapy >30 Gy within 6 months of the first dose of study therapy
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Known central nervous system metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Had allogeneic tissue/solid organ transplantation
* Interstitial lung disease or history of pneumonitis that has required oral or IV steroids
* Has received or will receive a live vaccine within 30 days prior to the first study therapy (seasonal flu vaccines that do not contain live vaccine are permitted)
* Active infection requiring intravenous systemic therapy
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or C
* Regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wu YL, Zhang L, Fan Y, Zhou J, Zhang L, Zhou Q, Li W, Hu C, Chen G, Zhang X, Zhou C, Dang T, Sadowski S, Kush DA, Zhou Y, Li B, Mok T. Randomized clinical trial of pembrolizumab vs chemotherapy for previously untreated Chinese patients with PD-L1-positive locally advanced or metastatic non-small-cell lung cancer: KEYNOTE-042 China Study. Int J Cancer. 2021 May 1;148(9):2313-2320. doi: 10.1002/ijc.33399. Epub 2020 Dec 9. PMID 33231285
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The China extension study enrolled 262 participants. Of the 262 total participants enrolled, 92 were previously enrolled in the global study for MK-3475-042 (NCT02220894).
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg by IV infusion on Day 1 every 3 weeks (Q3W) for a maximum of 35 cycles (21-day cycles). Participants who stopped the initial course of pembrolizumab due to complete response or had completed the initial course of pembrolizumab and had stable disease, but progressed after discontinuation, were eligible for a second course of pembrolizumab for up to an additional 1 year (17 additional 21-day cycles).
- Chemotherapy (SOC Treatment): Participants received carboplatin at target dose Area Under the Curve (AUC 5) (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + paclitaxel 200 mg/m^2 by IV infusion on Day 1 Q3W for a maximum of 6 cycles (21-day cycles) OR carboplatin target dose AUC 5 (maximum dose 750 mg) or AUC 6 (maximum dose 900 mg) + pemetrexed 500 mg/m^2 by IV infusion on Day 1 Q3W for a maximum of 6 cycles (21-day cycles). Participants with non-squamous histologies received optional additional maintenance treatment with pemetrexed 500 mg/m^2 by IV infusion on Day 1 Q3W.
Period: Overall Study
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Started | 128 | 134
Treated | 128 | 125
Received Second Course of Pembrolizumab | 5 | 0
Completed | 0 | 0
Not Completed | 128 | 134
Not completed — Adverse Event | 16 | 10
Not completed — Death | 87 | 107
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Participation in study terminated by Sponsor | 23 | 11

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment) | Total
Number analyzed (Participants) | 128 | 134 | 262
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (8.1) | 61.5 (8.0) | 61.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 105 | 119 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 128 | 134 | 262
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 128 | 134 | 262
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature; Grade 2: Ambulatory & capable of all selfcare but unable to carry out any work activities, up & about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled, cannot carry on any selfcare, totally confined to bed or chair or Grade 5: Dead.
  Participants
    ECOG PS=0 | 31 | 29 | 60
    ECOG PS=1 | 97 | 105 | 202
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Expression Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression status by immunohistochemistry assay using tumor tissue from an archival or newly obtained biopsy. Participants with a tumor proportion score (TPS) were classified as follows: ≥50% = PD-L1 strongly positive; 1-49% = PD-L1 weakly positive; and <1% = PD-L1 negative.
  Participants
    TPS=≥50% | 72 | 74 | 146
    TPS=20-49% | 29 | 29 | 58
    TPS=1-19% | 27 | 31 | 58
    TPS=<1% | 0 | 0 | 0
Tumor Histology [Count of Participants; unit: Participants] — Participants were classified according to tumor histology: Squamous or Non-squamous. The tumor histology determined potential treatment regimen.
  Participants
    Squamous | 71 | 76 | 147
    Non-squamous | 57 | 58 | 115

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With a Tumor Proportion Score (TPS) of ≥50%
Description: OS was determined for participants with a TPS of ≥50% and was defined as the time from randomization until death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. The OS for participants with a TPS ≥50% is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥50%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 72 | 74
Months | 20.0 [15.5 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 14.0 [10.0 to 17.9]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.38 to 1.00] — Hazard ratio based on Cox regression model with treatment as a covariate stratified by ECOG PS (0 vs. 1), and histology (squamous vs. non-squamous)

2. Primary Outcome: Overall Survival (OS) in Participants With a Tumor Proportion Score (TPS) of ≥20%
Description: OS was determined for participants with a TPS of ≥20% and was defined as the time from randomization until death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. The OS for participants with a TPS ≥20% is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥20%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 101 | 103
Months | 20.0 [17.4 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 13.7 [10.1 to 17.9]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.41 to 0.95] — Hazard ratio based on Cox regression model with treatment as a covariate stratified by ECOG PS (0 vs. 1), PD-L1 expression status (TPS=≥50% vs. TPS=1-49%), and histology (squamous vs. non-squamous)

3. Primary Outcome: Overall Survival (OS) in Participants With a Tumor Proportion Score (TPS) of ≥1%
Description: OS was determined for participants with a TPS of ≥1% and was defined as the time from randomization until death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data. The OS for participants with a TPS ≥1% is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥1%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 128 | 134
Months | 20.0 [17.4 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 13.7 [10.1 to 17.9]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.45 to 0.94] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥50%
Description: PFS was determined for participants with a TPS of ≥50% and was defined as the time from randomization until the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions or progression in non-target lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data. The PFS for participants with a TPS ≥50% is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥50%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 72 | 74
Months | 8.3 [4.2 to 10.6] | 6.5 [4.4 to 9.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.57 to 1.28] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥20%
Description: PFS was determined for participants with a TPS of ≥20% and was defined as the time from randomization until the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions or progression in non-target lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data. The PFS for participants with a TPS ≥20% is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥20%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 101 | 103
Months | 6.3 [4.2 to 8.4] | 6.5 [5.9 to 8.5]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.70 to 1.39] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥1%
Description: PFS was determined for participants with a TPS of ≥1% and was defined as the time from randomization until the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions or progression in non-target lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data. The PFS for participants with a TPS ≥1% is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥1%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 128 | 134
Months | 6.3 [4.2 to 8.3] | 6.4 [5.9 to 7.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.74 to 1.35] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥50%
Description: ORR was determined for participants with a TPS of ≥50%. ORR was determined per RECIST 1.1 and was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target and non-target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The percentage of participants who had a TPS ≥50% and who experienced a CR or PR is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥50%.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 72 | 74
Percentage of participants | 41.7 [30.2 to 53.9] | 24.3 [15.1 to 35.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Stratified Miettinen and Nurminen; Difference in Percentage (DP) = 17.2, 95% CI 2-sided [1.8 to 31.6] — DP for pembrolizumab vs. chemotherapy based on Miettinen & Nurminen method stratified by ECOG PS (0 vs. 1) and histology (squamous vs. non-squamous)

8. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥20%
Description: ORR was determined for participants with a TPS of ≥20%. ORR was determined per RECIST 1.1 and was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target and non-target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The percentage of participants who had a TPS ≥20% and who experienced a CR or PR is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥20%.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 101 | 103
Percentage of participants | 35.6 [26.4 to 45.8] | 24.3 [16.4 to 33.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Difference in Percentage (DP) = 11.3, 95% CI 2-sided [-1.4 to 23.7] — DP for pembrolizumab vs. chemotherapy based on Miettinen & Nurminen method stratified by ECOG PS (0 vs. 1), PD-L1 expression status (TPS=≥50% vs. TPS=1-49%), and histology (squamous vs. non-squamous)

9. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With a Tumor Proportion Score (TPS) of ≥1%
Description: ORR was determined for participants with a TPS of ≥1%. ORR was determined per RECIST 1.1 and was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target and non-target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The percentage of participants who had a TPS ≥1% and who experienced a CR or PR is presented.
Time Frame: Up to 23.2 months
Population: The analysis population included all participants who were alive at the time of randomization and had a TPS of ≥1%.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 128 | 134
Percentage of participants | 32.8 [24.8 to 41.7] | 24.6 [17.6 to 32.8]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy (SOC Treatment); Test type: Other; Difference in Percentage (DP) = 8.0, 95% CI 2-sided [-3.0 to 18.9] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: Up to 59.7 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 128 | 125
Participants | 126 | 124

11. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to 56.7 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment)
Number analyzed (Participants) | 128 | 125
Participants | 26 | 22

ADVERSE EVENTS:
Time Frame: Up to 70.4 months
Description: All-cause mortality=all randomized participants. Adverse events (AEs)=all participants who received ≥1 dose of treatment. Per protocol, disease progression was not considered an AE unless related to treatment. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression, malignant neoplasm progression, and disease progression not related to treatment were excluded.
Groups:
- Pembrolizumab Second Course: Participants who met the criteria for a second course of pembrolizumab received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle for up to an additional 1 year (17 additional 21-day cycles) of treatment.
Arm/Group | Pembrolizumab | Chemotherapy (SOC Treatment) | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 99/128 | 117/134 | 4/5
Serious Adverse Events (participants affected / at risk) | 42/128 | 41/125 | 2/5
Other Adverse Events (participants affected / at risk) | 119/128 | 119/125 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=128) | Chemotherapy (SOC Treatment) (N=125) | Pembrolizumab Second Course (N=5)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9) | 11 (13) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=128) | Chemotherapy (SOC Treatment) (N=125) | Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 39 (49) | 72 (116) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 16 (46) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 15 (27) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 7 (10) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 7 (9) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 15 (18) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 8 (9) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 7 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 17 (19) | 30 (37) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (19) | 13 (15) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (12) | 24 (36) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (11) | 18 (23) | 1 (1)
Asthenia (General disorders) | 6 (7) | 10 (11) | 0 (0)
Chest discomfort (General disorders) | 7 (8) | 7 (8) | 0 (0)
Chest pain (General disorders) | 6 (8) | 15 (16) | 1 (1)
Fatigue (General disorders) | 10 (13) | 20 (38) | 0 (0)
Malaise (General disorders) | 7 (7) | 18 (19) | 0 (0)
Pyrexia (General disorders) | 29 (42) | 23 (24) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (18) | 4 (8) | 0 (0)
Pneumonia (Infections and infestations) | 10 (12) | 6 (7) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 19 (24) | 11 (12) | 0 (0)
Alanine aminotransferase increased (Investigations) | 28 (47) | 31 (55) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 27 (39) | 26 (44) | 1 (1)
Bilirubin conjugated increased (Investigations) | 10 (13) | 4 (9) | 0 (0)
Blood albumin decreased (Investigations) | 4 (5) | 8 (9) | 0 (0)
Blood bilirubin increased (Investigations) | 13 (16) | 7 (9) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 8 (9) | 4 (9) | 0 (0)
Blood urea increased (Investigations) | 8 (9) | 2 (2) | 0 (0)
Blood uric acid increased (Investigations) | 7 (8) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 14 (19) | 11 (25) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (4) | 69 (232) | 0 (0)
Platelet count decreased (Investigations) | 5 (10) | 29 (87) | 1 (1)
Weight decreased (Investigations) | 18 (20) | 15 (19) | 2 (2)
White blood cell count decreased (Investigations) | 4 (5) | 64 (241) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 24 (25) | 38 (66) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (16) | 7 (9) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 12 (20) | 6 (21) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (23) | 19 (28) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 11 (13) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (25) | 11 (16) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (31) | 13 (18) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 12 (17) | 11 (19) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (34) | 15 (25) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (22) | 9 (10) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (13) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9) | 13 (16) | 0 (0)
Dizziness (Nervous system disorders) | 8 (9) | 5 (5) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 11 (13) | 0 (0)
Insomnia (Psychiatric disorders) | 14 (19) | 14 (25) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (36) | 19 (19) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 17 (17) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 11 (12) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 7 (7) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 32 (33) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (29) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 23 (26) | 6 (7) | 0 (0)
Hypertension (Vascular disorders) | 5 (8) | 7 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT03850444/Prot_SAP_001.pdf